CLINICAL TRIAL: NCT01146314
Title: A Family Based Intervention to Reduce the Risk of Type 2 Diabetes in Children
Acronym: FBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Principal Investigator, Amanda Lochrie, Principal Investigator, Nemours Children's Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-06038-001; 1-06-JF-33 (Other Grant/Funding Number: American Diabetes Association)
Record Dates: First submitted 2010-06-16; First posted 2010-06-17 (Estimated); Last update posted 2013-05-01 (Estimated); Status verified 2013-04

CONDITIONS: Pediatric Obesity; Type 2 Diabetes; Metabolic Syndrome
Keywords: family-focused intervention; pediatric obesity; diabetes prevention
MeSH Terms: conditions — Pediatric Obesity; Diabetes Mellitus, Type 2; Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lifestyle intervention (Experimental): A 6-month 14 session lifestyle intervention led by a psychologist and a dietitian for 90 minutes group sessions. Intervention sessions were help weekly, biweekly, and monthly over the course of 6 months.
  Interventions: Behavioral: Family Focused Lifestyle Intervention

INTERVENTIONS:
Behavioral: Family Focused Lifestyle Intervention — The lifestyle intervention is a 6-month intervention study lasting 6 months. The intervention is 14 sessions and conducted by a dietician and psychologist in a group setting with each intervention session lasting 90 minutes. The sessions are conducted weekly, biweekly, and monthly over the course of 6 months.

SUMMARY:
The purpose of this study was to determine if a family-focused lifestyle intervention helps to improve the health status, behaviors, and adjustment of overweight children.

DETAILED DESCRIPTION:
Type 2 diabetes (DM2), and obesity is increasing dramatically in the United States and worldwide among children. Even before children are diagnosed with DM2, they often show signs such as being overweight, having high blood pressure, abnormal lipid metabolism, and impaired glucose tolerance that put them at risk for other diseases, such as heart disease. In addition, children who are at risk for DM2 also face elevated risks of other major medical complications along with psychological and social consequences (e.g., depression, teasing, discrimination, school problems), which can often be just as damaging as the medical problems. Since obesity plays an important role in the progression to DM2, the need to prevent children from progressing to a diagnosis of DM2 is critical.

The proposed study was a randomized controlled trial comparing an education group for families of children at high risk for progression to metabolic syndrome and type 2 diabetes with a family-focused multi-component lifestyle intervention. The study addressed these specific aims:

1. Evaluated the effects of a family-focused lifestyle intervention on the health status of children at risk of metabolic syndrome (BMI, blood pressure, cholesterol, impaired glucose tolerance, waist circumference).
2. Evaluated the effects of a family focused psychosocial treatment on the health behaviors of children at risk for developing metabolic syndrome (eating behaviors, physical activity).
3. Evaluated the effects of a family focused psychosocial treatment on psychological outcomes of children at risk of developing metabolic syndrome (overall behavioral functioning, perception, self esteem, depression, quality of life).
4. Analyzed variables that are predictive of maintenance or termination of engagement in the family-focused lifestyle intervention.

It was hypothesized that this intervention approach will result in: a) improved health status and a reduction of risk for developing metabolic syndrome (BMI, waist circumference, blood pressure, cholesterol, and glucose levels), b) improved health behaviors (physical activity, diet), and c) generalize to more optimal psychosocial functioning (depression, self-perception, quality of life, school attendance) at short and long-term follow-up of the children in the intervention group compared with children in the education group.

ELIGIBILITY:
Inclusion Criteria:

* BMI 85th percentile and above, otherwise healthy
* Age between 8-11 years old

Exclusion Criteria:

* Diagnosis of metabolic syndrome
* Diagnosis of type 2 diabetes
* Diagnosis of Mental Retardation

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2006-09; Primary Completion 2009-12 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Improvement of health status of overweight children | Measured at 6 and 12 months
  Evaluated the effects of the intervention on improving BMI, blood pressure, waist circumference, and reducing the risk of the development of type 2 diabetes and metabolic syndrome.

SECONDARY OUTCOMES:
Improvement of health behaviors and psychosocial adjustment | Measured at 6 and 12 months
  Evaluated the effects of the intervention on changing health behaviors, such as eating patterns, diet, and eating behavior, and evaluate the effects of maintaining of improving adjustment to psychological stressors associated with being overweight (self esteem, depression, behavior).

CONTACTS AND LOCATIONS:
Overall Officials: Amanda S Lochrie, PhD, Principal Investigator — Nemours Children's Clinic
Locations (1):
- Nemours Children's Clinic, Jacksonville, Florida, United States

REFERENCES:
- [Derived] Kahhan N, Hossain MJ, Lang J, Harrison C, Canas J, Wysocki T, Lochrie A, Balagopal PB. Durability of Changes in Biomarkers of Cardiometabolic Disease: 1-Year Family-Based Intervention in Children with Obesity. Metab Syndr Relat Disord. 2021 Jun;19(5):264-271. doi: 10.1089/met.2020.0097. Epub 2021 Mar 1. PMID 33650888